CLINICAL TRIAL: NCT00874445
Title: Prospective Comparison of 50/50% Tilt and Tuned Defibrillation Waveforms in a Single Coil Active Can Configuration
Brief Title: Comparison of 50% Tilt and Tuned Waveforms in Single-Coil Active Can Configuration
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD 475
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICD shocks programmed to Tuned Waveform: ICD shocks programmed to Tuned Waveform
  Interventions: Device: ICD/ CRT-D
- ICD shocks programmed to Fixed Tilt Waveform: ICD shocks programmed to Fixed Tilt Waveform
  Interventions: Device: ICD/ CRT-D

INTERVENTIONS:
Device: ICD/ CRT-D — Patients in experimental group will have their ICDs programmed to Tuned waveform and those in the control group will have their ICDs programmed to Fixed Tilt waveform.

SUMMARY:
The purpose of this study is to compare the defibrillation efficacy between the 50/50% tilt biphasic waveform and the Tuned biphasic waveform in a single coil active can configuration.

DETAILED DESCRIPTION:
There has been one prospective study that found some benefit of using tuned waveforms over 50/50% tilt waveforms.11 Other studies have failed to show much change in defibrillation efficacy with different duration biphasic waveforms. A vast majority of patients in these studies were tested with dual coil leads. Although dual coil leads can lower defibrillation thresholds, it is known that dual coil leads can make the lead extraction difficult, lead to venous obstruction and are more prone to failure. Results from a recent study showed that that a single coil configuration is adequate in a vast majority of patients when DFT testing was performed with tuned waveforms. This makes the use of single-coil leads during ICD/ CRT-D implants an attractive option.

Theoretical analysis has shown that difference between the tuned and 50% tilt waveforms is amplified at high impedance levels with tuned waveforms being superior (unpublished). Accordingly, this study has been designed to prospectively compare the DFT estimates with tuned and 50% tilt waveforms in left-sided, active pectoral defibrillation lead systems when the SVC coil has been turned OFF or is not part of the shocking circuit.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets standard indication for an ICD/ CRT-D and will be implanted with an FDA approved SJM ICD/ CRT-D and compatible defibrillation lead system in the left pectoral region.
* Patient is able to tolerate DFT testing.

Exclusion Criteria:

* Patient has the pulse generator on the right side.
* Patient is pregnant.
* Patient is less than 18 years old.
* SVC coil was turned ON during DFT testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ICD/CRT-D indications
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
True DFTs in fixed tilt and tuned waveforms obtained in volts (V) | Implant

SECONDARY OUTCOMES:
True DFTs in fixed tilt and tuned waveforms obtained in joules (J) | Implant

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Michael Gold, Charleston, South Carolina, United States

REFERENCES:
- [Background] Gold M, Val-Mejias J, Leman RB, Tummala R, Goyal S, Kluger J, Kroll M, Oza A. Optimization of superior vena cava coil position and usage for transvenous defibrillation. Heart Rhythm. 2008 Mar;5(3):394-9. doi: 10.1016/j.hrthm.2007.12.001. Epub 2007 Dec 5. PMID 18313597
- [Background] Natarajan S, Henthorn R, Burroughs J, Esberg D, Zweibel S, Ross T, Kroll M, Gianola D, Oza A. "Tuned" defibrillation waveforms outperform 50/50% tilt defibrillation waveforms: a randomized multi-center study. Pacing Clin Electrophysiol. 2007 Jan;30 Suppl 1:S139-42. doi: 10.1111/j.1540-8159.2007.00624.x. PMID 17302691
- [Background] Mouchawar G, Kroll M, Val-Mejias JE, Schwartzman D, McKenzie J, Fitzgerald D, Prater S, Katcher M, Fain E, Syed Z. ICD waveform optimization: a randomized, prospective, pair-sampled multicenter study. Pacing Clin Electrophysiol. 2000 Nov;23(11 Pt 2):1992-5. doi: 10.1111/j.1540-8159.2000.tb07070.x. PMID 11139975
- [Result] Gold MR, Val-Mejias J, Cuoco F, Siddiqui M. Comparison of fixed tilt and tuned defibrillation waveforms: the PROMISE study. J Cardiovasc Electrophysiol. 2013 Mar;24(3):323-7. doi: 10.1111/jce.12041. Epub 2012 Dec 4. PMID 23210764
- [Derived] Gold MR, Yu Y, Singh JP, Birgersdotter-Green U, Stein KM, Wold N, Meyer TE, Ellenbogen KA. Effect of Interventricular Electrical Delay on Atrioventricular Optimization for Cardiac Resynchronization Therapy. Circ Arrhythm Electrophysiol. 2018 Aug;11(8):e006055. doi: 10.1161/CIRCEP.117.006055. PMID 30354310